CLINICAL TRIAL: NCT03437369
Title: Efficacy and Safety on Heart Rate Control With Ivabradine on Cardiogenic Shock (ES-FISH)
Brief Title: Efficacy and Safety on Heart Rate Control With Ivabradine on Cardiogenic Shock
Acronym: ES-FISH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Marcelo Sanmartín Fernández, Director Acute Coronary Syndrome Process, Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HURamonyCajal
Record Dates: First submitted 2018-01-15; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Cardiogenic Shock
Keywords: Ivabradine, heart rate, acute heart failure
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ivabradine (Experimental): Drug: Ivabradine Oral tablets 2.5 mg Dose: 10-15 mg/day Duration: 30 days
  Interventions: Drug: Ivabradine Oral Tablet
- Standard of Care (Other): The study drug will be compared with standard of Care treatment
  Interventions: Other: Standard of Care treatment

INTERVENTIONS:
Drug: Ivabradine Oral Tablet — The target dose is 10 to 15 mg / day, administered orally in two doses
  Arms: Ivabradine
Other: Standard of Care treatment — The study drug will be compared with the standard of Care treatment
  Arms: Standard of Care

SUMMARY:
This is a randomized 1:1 blinded study that evaluate in acute left heart failure-cardiogenic shock patients if ivabradine treatment can reduce pulmonary wedge pressure, without inducing a significant or relevant reduction in cardiac output or increasing the risk of arterial hypotension and with the benefit of allowing a faster titration of heart failure drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years, with acute heart failure due to left ventricular systolic dysfunction (LVEF ≤ 40%) in sinus rhythm, baseline HR ≥ 90 bpm, with signs of low peripheral perfusion with indication for intravenous inotropic treatment (catecholamines: dobutamine , adrenaline, dopamine or noradrenaline) and admitted to the Cardiological Intensive Care Unit.
* Pharmacological treatment and stable hemodynamic situation in the 4 hours before inclusion.
* Pulmonary wedge pressure ≥ 18 mm Hg and systolic blood pressure > 90 mm Hg.
* Patient's signature on the consent form.

Exclusion Criteria:

* Previous treatment with ivabradine (< 48 hours).
* Known hypersensitivity to ivabradine.
* Cardiac rhythm different from sinus rhythm.
* Unstable cardiac rhythm due to paroxysmal atrial fibrillation or atrial flutter, very frequent ventricular or supraventricular premature beats, ventricular tachycardia, 2nd or 3rd degree atrioventricular (AV) block.
* Severe chronic renal failure (estimated glomerular filtration rate ≤15 ml / min) or on chronic treatment with dialysis.
* QT interval higher than 450 ms.
* Sepsis as a probable mechanism of tachycardia and hypotension.
* Need for urgent cardiac surgery, planned within 72 hours of possible inclusion.
* Severe aortic stenosis or severe valvular disease that requires surgical correction.
* Patient must not have received an IV bolus of furosemide immediately before the baseline hemodynamic assessment.
* Severe hepatic insufficiency.
* Patient must not be participating in another clinical trial.
* Concomitant use of potent CYP3A4 inhibitors.
* Acute anemia or hypovolemia uncorrected.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in pulmonary wedge pressure and cardiac output after 24h-treatment with ivabradine or standard of care treatment. | 24 hours
  Reduction of pulmonary wedge pressure from baseline in both treatment arms (ivabradine arm versus standard of care treatment measured by Swan Ganz balloon flotation catheter)

SECONDARY OUTCOMES:
Severe bradycardia | 24 hours
  -Development of excessive bradycardia defined as heart rate (HR) <50 beats per minute
Arrhythmias | 24 hours
  New-onset of ventricular arrhythmias or atrial fibrillation
Hypotension | 24 hours
  Hypotension, defined as systolic blood pressure <90 mmHg
Time to withdrawal of vasoactive drugs | 30 days
  -Time to catecholamine withdrawal in both treatment arms (days)
Time needing invasive mechanical ventilation | 30 days
  Mechanical (invasive) ventilation time after initiation of ivabradine/control treatment.
B-type natriuretic peptide (BNP) | 30 days
  Measured B-type natriuretic peptide (BNP) values at 30 days
Left ventricular ejection fraction | 30 days
  Change in left ventricle ejection fraction from baseline in both treatment arms (%)
Cardiovascular mortality | 30 days
  Mortality due to cardiovascular causes
Total mortality | 30 days
  Mortality from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Sanmartín Fernández, PhD, Principal Investigator — Hospital Universitario Ramon y Cajal
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tardif JC, Ford I, Tendera M, Bourassa MG, Fox K; INITIATIVE Investigators. Efficacy of ivabradine, a new selective I(f) inhibitor, compared with atenolol in patients with chronic stable angina. Eur Heart J. 2005 Dec;26(23):2529-36. doi: 10.1093/eurheartj/ehi586. Epub 2005 Oct 7. PMID 16214830
- [Background] Swedberg K, Komajda M, Bohm M, Borer JS, Ford I, Dubost-Brama A, Lerebours G, Tavazzi L; SHIFT Investigators. Ivabradine and outcomes in chronic heart failure (SHIFT): a randomised placebo-controlled study. Lancet. 2010 Sep 11;376(9744):875-85. doi: 10.1016/S0140-6736(10)61198-1. PMID 20801500
- [Background] Fasullo S, Cannizzaro S, Maringhini G, Ganci F, Giambanco F, Vitale G, Pinto V, Migliore G, Torres D, Sarullo FM, Paterna S, Di Pasquale P. Comparison of ivabradine versus metoprolol in early phases of reperfused anterior myocardial infarction with impaired left ventricular function: preliminary findings. J Card Fail. 2009 Dec;15(10):856-63. doi: 10.1016/j.cardfail.2009.05.013. Epub 2009 Jul 3. PMID 19944362
- [Background] Lechat P, Hulot JS, Escolano S, Mallet A, Leizorovicz A, Werhlen-Grandjean M, Pochmalicki G, Dargie H. Heart rate and cardiac rhythm relationships with bisoprolol benefit in chronic heart failure in CIBIS II Trial. Circulation. 2001 Mar 13;103(10):1428-33. doi: 10.1161/01.cir.103.10.1428. PMID 11245648